CLINICAL TRIAL: NCT01768689
Title: The Effect of Active Adherence-Encouraging Interventions on Adherence to Tyrosine Kinase Inhibitor Treatment in Chronic Myeloid Leukemia - A Prospective Observational Multicenter Study (TAKE-IT)
Brief Title: Interventional Study to Improve Adherence to Tyrosine Kinase Inhibitors in Chronic Myeloid Leukemia
Acronym: TAKE-IT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: pia raanani (Other)
Responsible Party: Sponsor-Investigator, pia raanani, Prof. Pia Raanani, Rabin Medical Center
Organization: Rabin Medical Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TAKE IT - CML adherence
Record Dates: First submitted 2013-01-08; First posted 2013-01-15 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Medication Adherence
Keywords: adherence; chronic myeloid leukemia; tyrosine kinase inhibitors
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Medication Adherence

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: The adherence assessed per study protocol was masked to participants and care providers during the preintervention and post intervention phases. At the time of intervention participants were notified once of their adherence as part of the feedback-based intervention
Oversight: Data Monitoring Committee: No

ARMS (2):
- Run-in period (No Intervention): First 3 months of study during which adherence will be measured for each consecutively included study subject, but no intervention will be performed. Patient will receive routine treatment for CML according to the physician discretion.
- Adherence-encouraging period (Experimental): Months 4 to 9 of study during which adherence will be measured for each consecutively included study subject, while implementing adherence-encouraging interventions:
  1. adherence-encouraging interventions - Group meetings
  2. adherence-encouraging interventions - Individual meetings
  3. adherence-encouraging interventions - Monthly phone calls
  Patient will receive routine treatment for CML according to the physician discretion.
  Interventions: Behavioral: Adherence-encouraging interventions - Group meeting; Behavioral: Adherence-encouraging interventions - Individual meetings; Behavioral: Adherence-encouraging interventions - Monthly phone calls

INTERVENTIONS:
Behavioral: Adherence-encouraging interventions - Group meeting — One Group meeting (at the beginning of the intervention period) for all participants, focusing on issues relevant to adherence improvement
  Arms: Adherence-encouraging period
Behavioral: Adherence-encouraging interventions - Individual meetings — Individual meetings focusing on adherence issues with a multidiscilinary team
  Arms: Adherence-encouraging period
Behavioral: Adherence-encouraging interventions - Monthly phone calls — Monthly phone calls to detect urgent adherence-related issues
  Arms: Adherence-encouraging period

SUMMARY:
Adherence to tyrosine kinase inhibitors is associated with improved outcomes in chronic myeloid leukemia patients. Hence, improved adherence might improve CML patients' prognosis.

Decreased adherence is a common problem in such patients, with non-adherence in up to 30% of patients in several studies. Recently, an emphasis has been placed on improving patient's adherence to tyrosine kinase inhibitors in these patients. However, there is no prospective high-quality evidence showing that adherence can be improved in these patients.

Therefore, the investigators hypothesize that adherence-encouraging interventions improve adherence to tyrosine kinase inhibitors in chronic myeloid leukemia patients.

DETAILED DESCRIPTION:
The cytogenetic hallmark of chronic myeloid leukemia (CML) is the reciprocal translocation between chromosomes 9 and 22 creating the Philadelphia (Ph(1)) chromosome. The BCRABL1 fusion gene is the result of this translocation and encodes for a constitutively active tyrosine kinase responsible for the development of CML. Tyrosine kinase inhibitors (TKIs) targeting the protein product of this aberrant gene, the BCRABL-1 protein, have revolutionized the therapeutic approach to chronic myeloid leukemia (CML). Treatment with the first FDA approved TKI, imatinib mesylate (Gleevec, Novartis), in chronic phase CML results in a projected 8 year overall survival of 85%. Recently, two second generation TKIs, Dasatinib and Nilotinib, have been approved for use in newly diagnosed chronic phase CML, as a result of studies showing improved molecular and cytogenetic outcomes. Importantly, in each of the above studies there was a substantial number of dropouts due to drug intolerance and resistance, among other reasons. In a prospective observational study of 169 CML patients, only 14% of patients were fully adherent with prescribed imatinib. Moreover, one third of patients were considered to be non-adherent, which is similar to the proportion of dropouts in the landmark studies on TKIs in CML. Thus, it is clear that there is a subgroup of patients who do not properly adhere to treatment. This is especially significant because the contemporary approach to CML in complete cytogenetic remission (CCyR) and major molecular remission (MMR) necessitates long-term, chronic treatment with TKIs.

Therefore, although hematologists have the luxury of an armamentarium of highly effective drugs, one of the most challenging aspects of treating CML is the management of non-compliance to TKI treatment. TKI-induced adverse effects are only one of a wide spectrum of reasons for non-adherence to TKI treatment.

Recently several studies have demonstrated the prognostic importance of adhering to imatinib treatment. In a pivotal study of 87 chronic phase CML (CP-CML) patients in CCyR, an adherence rate of > 90% strongly correlated with the 6 year probability of achieving MMR (94.5% vs. 28.4% when adherence rates were ≤ 90%). Non-adherence to imatinib treatment also adversely affects event free survival and is associated with loss of CCyR in patients on long term treatment. These data support the intuitive concept that CML can be effectively treated with the drugs currently available, as long as patients adhere to treatment. Moreover, non-adherence to imatinib treatment has been associated with increased economic burden and healthcare costs. Consequently, TKI adherence is an attractive potential target for intervention.

Non-adherence to medication is an intricate problem that is influenced by the physician, the healthcare system, and economic and social factors. Other medical disciplines have assessed various modes of improving adherence to therapeutic regimens, with varying success. A recent study assessing adherence-related behavior among CML patients, demonstrated that among a multitude of reasons for non-adherence, patient forgetfulness and drug side effects were the most common causes of unintentional and intentional non-adherence, respectively. Several methods of improving adherence among patients with CML were retrospectively assessed by Moon et al. Subjects in the intervention arm were more likely to receive prescriptions for imatinib than those receiving standard care (98.2 ± 0.03% vs. 79.3 ± 0.16%). Although there was no difference in adherence to prescribed treatment between the two groups, the overall compliance, a composite endpoint of the above two outcomes, was markedly improved in the intervention group ((93.0 ± 2.3% vs. 76.2 ± 7.4%, P = 0.001). Recently, Gater et al conceived a conceptual model aimed at improving adherence in CML patients treated with 1st and 2nd generation TKIs, based on a systematic review of the literature. However, there are currently no prospective data evaluating whether adherence in CML can be influenced by active intervention.

Study Hypothesis:

Adherence to tyrosine kinase inhibitors (TKIs) is associated with improved outcomes in chronic myeloid leukemia (CML) patients. Hence, improved adherence might improve CML patients' prognosis.

The investigators hypothesize that adherence-encouraging interventions improve adherence to TKIs in CML patients.

Study Objective:

1. Primary Objective: By means of a prospective before-after study, the investigators aim to assess whether specific adherence-encouraging interventions improve TKI adherence in patients with CP-CML treated by these agents. The investigators will target previously documented reasons for non-adherence 11 with interventions that were selected based on prior experience in other medical disciplines and will evaluate their contribution to patients' adherence to treatment.
2. To better understand non-adherence in CML and pinpoint independent risk factors for non-adherence
3. To validate questionnaires assessing adherence, and evaluate whether they could be of use in indentifying patients at risk for non-adherence
4. To compare adherence to second generation TKIs with adherence to imatinib
5. To assess the role of a clinical pharmacist in preventing potential drug interactions
6. To determine whether the intervention has a long term effect on adherence during one year of post-intervention follow up
7. To estimate long term effects of adherence on clinical, cytogenetic and molecular outcomes

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic phase chronic myeloid leukemia (CP-CML), aged 18 years or older

  * CP-CML defined as: Medical history of cytogenetically confirmed CP-CML defined as the presence of the Philadelphia chromosome on bone marrow aspirates (a minimum of 20 metaphases is required; FISH cannot be used). If Philadelphia chromosome was negative or if cytogenetic results were not available, BCR-ABL-positive CML patients can be included.
* At least 3 months of TKI treatment (imatinib, dasatinib or nilotinib) before study initiation.

Exclusion Criteria:

* Current or prior accelerated/blast phase or stem cell transplant
* Participation in another interventional study
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Clinically relevant change in MEMS-measured adherence | From 3 months before intervention, until 3 months after starting the intervention
  Improvement in a patient's adherence from less than 90% during the initial 3 month run-in period, to 90% or more during the first 3 months of intervention.
  Definitions:
  1. Adherence above 90% was defined as clinically relevant.
  2. Adherence rate = actual calculated dose/prescribed dose.
  3. Adherence will be calculated from "medical events monitoring system" (MEMS) data which will be collected continuously throughout the first 7.5 months of the study period. MEMS is an electronic monitoring system designed to compile the dosing histories of ambulatory patients prescribed oral medications
General improvement in MEMS-measured adherence | 3 months prior to the intervention, until 3 months after starting the intervention
  An absolute improvement of 10% in a patient's adherence, between their adherence during the initial 3 month run-in period and their adherence during the first 3 months of intervention.
  See Definitions of adherence rate and measurement of adherence in the first primary outcome description.

SECONDARY OUTCOMES:
Mean-difference in MEMS-measured adherence | 3 months prior to intervention until 3 months after starting the intervention
  Mean-difference in adherence (as measured by the MEMS) between the run-in period and the first 3 months of the intervention period (paired t-test).
  The aim is to evaluate whether such a difference exists and whether it has statistical significance.
  For more details on the MEMS system, please see the description under the primary outcome.
Mean change in The Basel Assessment of Adherence to Tyrosine Kinase Inhibitors Scale (BAATIS) | 1) Short term: 3 months prior to intervention until 6 months after starting the intervention; 2) Long term: 3 months prior to intervention until 18 months after starting the intervention
  Mean-difference in BAATIS scale scores between the run-in period and the intervention period (paired t-test)
  The BAATIS is a clinician reported outcome which has been used to assess adherence to immunosuppressive medication in solid organ transplant patients (BAASIS; Basal assessment of adherence with the Immunosuppressive Regimen Scale). Noens et al adapted the questionnaire for use among CML patients in the ADAGIO study. We have performed a similar adaptation
  Regarding time frames:
  Each questionnaire-related secondary outcome will be evaluated at two time frames:
  1. Short term, to assess an immediate effect on adherence
  2. Long term follow up (up to one year after the end of the intervention period) in order to determine whether the intervention has a long term effect on adherence.
Effect of intervention on tyrosine kinase inhibtor related adverse events | 3 months prior to intervention until 6 months after starting the intervention
  The incidence of tyrosine kinase inhibitor related adverse events during 6 months of intervention compared to that witnessed during the initial 3 month run-in period
Adverse effects of tyrosine kinase inhibitors as a measure of MEMS-measured adherence | 3 months prior to intervention until 3 months after starting the intervention
  The incidence of tyrosine kinase inhibtor related adverse events throughout the first 6 months of the study period as a function of adherence (measured by MEMS)
Percentage of patients improving in patient self-reported non-adherence | 3 months prior to intervention until 6 months after starting the intervention
  The percentage of patients changing from a self-reported non-adherence of "yes" during the run-in period, to a self-reported non-adherence of "no" after the intervention, compared to the percentage of those who answered "yes" during the study period and remained "yes" after the intervention.
  Definition of the "Patient self-reported question regarding non-adherence":
  Each patient is asked the following question:
  "It is common that patients at times miss a few doses, for a whole range of reasons. Thinking of the past 7 days have you missed any doses?"
  If a patient answers 'yes' it will be taken as an indication that the patient has problems with adherence.
Mean change in the physician visual analogue scale (VAS) of adherence | 1) Short term: 3 months prior to intervention until 6 months after starting the intervention; 2) Long term: 3 months prior to intervention until 18 months after starting the intervention
  Mean-difference in physician visual analogue scale (VAS) of adherence scores between the run-in period and the intervention period (paired t-test).
  The physician VAS on adherence rates patient adherence (as assessed by a physician) on a 10 cm VAS scale. A similar scale is in widespread use in several clinical disciplines, especially in assessing pain. It has also been used in assessing adherence to medication.
  The VAS ranges from perfect adherence (100% = 100mm) to no adherence (0% = 0mm).
  Regarding time frames:
  Each questionnaire-related secondary outcome will be evaluated at two time frames:
  1. Short term, to assess an immediate effect on adherence
  2. Long term follow up (up to one year after the end of the intervention period) in order to determine whether the intervention has a long term effect on adherence.
Mean change in the patient visual analogue scale (VAS) of adherence | 1) Short term: 3 months prior to intervention until 6 months after starting the intervention; 2) Long term: 3 months prior to intervention until 18 months after starting the intervention
  Mean-difference in patient visual analogue scale (VAS) of adherence scores between the run-in period and the intervention period (paired t-test).
  The patient VAS on adherence rates patient adherence (as assessed by the patient) on a 10 cm VAS scale.
  See detailed explanation on the VAS under the outcome "Mean change in the physician visual analogue scale (VAS) of adherence"
  Regarding time frames:
  Each questionnaire-related secondary outcome will be evaluated at two time frames:
  1. Short term, to assess an immediate effect on adherence
  2. Long term follow up (up to one year after the end of the intervention period) in order to determine whether the intervention has a long term effect on adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Pia Raanani, MD, Principal Investigator — Rabin Medical Center
Locations (4):
- Israel (4):
  - Soroka Medical Center, Beersheba
  - Rambam Medical Center, Haifa
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Petah Tikva

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Noens L, van Lierde MA, De Bock R, Verhoef G, Zachee P, Berneman Z, Martiat P, Mineur P, Van Eygen K, MacDonald K, De Geest S, Albrecht T, Abraham I. Prevalence, determinants, and outcomes of nonadherence to imatinib therapy in patients with chronic myeloid leukemia: the ADAGIO study. Blood. 2009 May 28;113(22):5401-11. doi: 10.1182/blood-2008-12-196543. Epub 2009 Apr 6. PMID 19349618
- [Background] Eliasson L, Clifford S, Barber N, Marin D. Exploring chronic myeloid leukemia patients' reasons for not adhering to the oral anticancer drug imatinib as prescribed. Leuk Res. 2011 May;35(5):626-30. doi: 10.1016/j.leukres.2010.10.017. Epub 2010 Nov 20. PMID 21095002
- [Background] Gater A, Heron L, Abetz-Webb L, Coombs J, Simmons J, Guilhot F, Rea D. Adherence to oral tyrosine kinase inhibitor therapies in chronic myeloid leukemia. Leuk Res. 2012 Jul;36(7):817-25. doi: 10.1016/j.leukres.2012.01.021. Epub 2012 Feb 23. PMID 22364811
- [Background] Marin D, Bazeos A, Mahon FX, Eliasson L, Milojkovic D, Bua M, Apperley JF, Szydlo R, Desai R, Kozlowski K, Paliompeis C, Latham V, Foroni L, Molimard M, Reid A, Rezvani K, de Lavallade H, Guallar C, Goldman J, Khorashad JS. Adherence is the critical factor for achieving molecular responses in patients with chronic myeloid leukemia who achieve complete cytogenetic responses on imatinib. J Clin Oncol. 2010 May 10;28(14):2381-8. doi: 10.1200/JCO.2009.26.3087. Epub 2010 Apr 12. PMID 20385986
- [Background] Osterberg L, Blaschke T. Adherence to medication. N Engl J Med. 2005 Aug 4;353(5):487-97. doi: 10.1056/NEJMra050100. No abstract available. PMID 16079372
- [Background] Moon JH, Sohn SK, Kim SN, Park SY, Yoon SS, Kim IH, Kim HJ, Kim YK, Min YH, Cheong JW, Kim JS, Jung CW, Kim DH. Patient counseling program to improve the compliance to imatinib in chronic myeloid leukemia patients. Med Oncol. 2012 Jun;29(2):1179-85. doi: 10.1007/s12032-011-9926-8. Epub 2011 Apr 7. PMID 21472487
- [Background] Jonsson S, Olsson B, Soderberg J, Wadenvik H. Good adherence to imatinib therapy among patients with chronic myeloid leukemia--a single-center observational study. Ann Hematol. 2012 May;91(5):679-685. doi: 10.1007/s00277-011-1359-0. Epub 2011 Nov 3. PMID 22048790